CLINICAL TRIAL: NCT06575426
Title: A Phase I/IIa, Single Site, Open-Label, Ascending Dose Study to Evaluate the Safety and Efficacy of OPF-310 [Encapsulated Porcine Islet Cells for Xenotransplantation] in Subjects With Type 1 Diabetes Mellitus
Brief Title: A Study to Investigate Safety and Effectiveness of Porcine Pancreatic Cells (OPF-310) in Patients With Type 1 Diabetes Mellitus
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Factory, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 215-001
Record Dates: First submitted 2024-08-20; First posted 2024-08-28 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 1; Hypoglycemia; Islet Cell Transplantation
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type1; T1DM; Hypoglycemia; islet cell transplantation; pig islet cell transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: A Phase I/IIa, Single site, Open-Label, Ascending Dose Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- OPF-310 (Experimental): 13 patients will be transplanted OPF-310.
  Interventions: Combination Product: OPF-310

INTERVENTIONS:
Combination Product: OPF-310 — Dose(Part1): 6,000 islet equivalents (IEQ)/kg or 12,000 islet equivalents (IEQ)/kg
  Dose(Part2): Recommended Phase II Dose(RP2D), which will be determined based on the data of Part1
  * In Part1, three subjects will be enrolled into the first dosing cohort (Cohort 1: 6,000 IEQ/kg) and they will undergo safety monitoring. Three subjects in Cohort 2 will be dosed with 12,000 IEQ/kg and will undergo safety monitoring.
  * In Part2, 7 subjects will be enrolled into the Part 2 dose-expansion part.

SUMMARY:
This study is First In Human study for Encapsulated Porcine Islet Cells for Xenotransplantation (OPF-310). The purpose of this study to assess the safety, tolerability, and efficacy of OPF-310 transplantation and to define the recommended Phase 2 dose (RP2D) in adult subjects with unstable Type 1 Diabetes Mellitus (T1DM) and a level 3 (severe) hypoglycemic episode at least three times within the 1 year prior to enrollment despite treatment with a closed loop system (CLS) for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be aged 35 to 65 years of age inclusive, at the time of signing the informed consent.
2. Subject has an established diagnosis of type 1 diabetes mellitus (T1DM)(in accordance with the American Diabetes Association's criteria), with a minimum duration since diagnosis of 5 years.
3. If one of the following criteria (either a or b) applies:

   1. Subject has unstable T1DM, not achieving adequate control after receiving CLS (CGM:Dexcom G6, insulin pump: Omnipod® 5 or t:slim X2) under care of a qualified diabetes team for at least 6 months prior to enrollment.
   2. Subject has unstable T1DM, not achieving adequate control after receiving CLS (CGM:Dexcom G7, insulin pump: Omnipod® 5, t:slim X2, iLet Bionic Pancreas or The Tandem Mobi System) under care of a qualified diabetes team for at least 6 months prior to enrollment.
4. If one of the following criteria (either a, b or c) applies:

   1. Subject has had a Level 3 (severe) hypoglycemic episode (defined as having cognitive impairment requiring external assistance for recovery) at least three times within the 1 year prior to enrollment recorded in the medical record or patient log.
   2. Subject has had a Level 3 (severe) hypoglycemic episode at least once within the 1 year prior to enrollment and demonstrates a Clarke Score ≥4, assessed by trained study personnel. The SHE(s) and Clarke Score must be recorded in the medical record or patient log.
   3. Subject has had TBR >1% at glucose levels below 70mg/dL and demonstrates a Clarke Score≥4, assessed by trained study personnel. TBR data used for screening and Clarke score must be recorded in the medical record or patient log.
5. Subject has C-peptide <0.3 ng/mL following a mixed meal tolerance test or undetectable fasting C-peptide.
6. Hemoglobin A1C (HbA1c) ≤ 9.0
7. Contraceptive use must be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
8. Subject who can agree to cooperate with lifetime follow-up after transplantation.
9. Subject is capable of providing signed informed consent

Exclusion Criteria:

1. Previous history of insulin resistance (defined as an average insulin dose requirement ≥ 0.8 unit/kg/day for 1 week prior to enrollment).
2. Subject has latent autoimmune diabetes in adults (LADA), ketosis-prone (Flatbush) diabetes, or maturity onset diabetes of the young (MODY).
3. CRP ≥ 10 mg/L.
4. Clinically unstable thyroid disease (thyroid stimulating hormone (TSH)< the lower limit of the normal range of TSH at the site.) Patients with subclinical hyperthyroidism can be rescreened once TSH levels normalize due to treatment or other factors. In addition, patients with transiently abnormal TSH levels may undergo rescreening only once during the screening period.
5. History of malignancies within the past 5 years, excluding basal and squamous cell carcinoma
6. Positive serologies or nucleic acid testing for human immunodeficiency virus (HIV), hepatitis C, and hepatitis B.
7. Active or untreated proliferative diabetic retinopathy. Subjects may be rescreened once they are successfully treated.
8. Serious comorbid conditions that are likely to affect participation in the study, including:

   1. Within the last 12 months, peripheral vascular disease with previous amputation.
   2. History of New York Heart Association (NYHA) class II, III or IV congestive heart failure (CHF) and/or chronic atrial fibrillation.
   3. Chronic obstructive pulmonary disease (COPD) or asthma with previous hospitalization for decompensation; a requirement for mechanical ventilation at any stage; or long- term treatment with oral corticosteroids.
   4. Macroalbuminuria (> 300 mg albumin/gm creatinine).
   5. Estimated glomerular filtration rate (eGFR) cut-off of < 30 ml/min for all per Kidney Disease Improving Global Outcomes (KDOQI) and Kidney Disease Outcomes Quality Initiative (KDIGO) consensus.
9. Use of warfarin or other anticoagulant therapy (except aspirin), or prothrombin time and international normalized ratio (PT-INR) > 1.5
10. Adrenal insufficiency being treated with corticosteroids
11. Previous pan-peritonitis
12. Previous cardiovascular or cerebrovascular disease
13. Patients with hematopoietic stem cell abnormalities (e.g., aplastic anemia, myelodysplastic syndrome)
14. Patients who received a blood transfusion in the previous 90 days, are anticipated to undergo surgery during the 1-year study period that may require transfusion, or have donated blood within the previous 90 days.
15. Previous receipt of an organ, skin allograft, or other tissue transplant from an allogeneic human or animal donor.
16. Treatment with immunosuppressive medication.
17. Previous abdominal surgery, excluding uncomplicated appendectomy, cholecystectomy, exploratory laparoscopy and hernia repair performed prior to 12 weeks prior to enrollment.
18. Treatment with any non-insulin hypoglycemic medication not intended to be used as an adjunct to insulin therapy.
19. Treatment with acetaminophen or hydroxycarbamide.
20. Use of any investigational products within 12 weeks of enrollment (before entering run-in) or 5 half-lives of the investigational product, whichever is greater.
21. Subject has history of allergy to antibiotics (Amphotericin B, Cefazolin, Ciprofloxacin, Gentamicin), which are used during manufacture of OPF-310.
22. Previous history of insulin allergy (including porcine insulin), pork product allergy or alginate/seaweed allergy.
23. Panel reactive antibodies (PRA) > 80 %.
24. Active drug, substance or alcohol addiction.
25. Body mass index (BMI) >27 kg/m2.
26. Any other condition that, in the opinion of the Investigator, may interfere with adherence to the study protocol, including dementia, psychiatric disorder, medical condition, or a history of non-adherence to appointments or treatments

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Subjects Reaching the Efficacy Goal | One year after transplant
  A successful primary endpoint was defined as achieve both an HbA1c < 7 % and a reduction of at least 0.5% from baseline, and absence of a Level 3 (severe) hypoglycemic episode from 12 weeks to 52 weeks post-transplant.

SECONDARY OUTCOMES:
Percentage reduction in nocturnal hypoglycemic event rate | 12 week, 24 week 52 weeks after transplant
  Change from baseline in nocturnal hypoglycemic event rate specified in the protocol
Percentage improvement in time below range (<70 mg/dl) by continuous glucose monitoring (CGM) | 12 week, 24 week 52 weeks after transplant
  Change from baseline in the CGM data specified in the protocol
Percentage improvement in time in range (70-180 mg/dl) by CGM | 12 week, 24 week 52 weeks after transplant
  Change from baseline in the CGM data specified in the protocol
Percentage improvement in time above range (>180 mg/dl) by CGM | 12 week, 24 week 52 weeks after transplant
  Change from baseline in the CGM data specified in the protocol
Change in mean amplitude of glycemic excursion (MAGE) by CGM. | 12 week, 24 week 52 weeks after transplant
  Change from baseline in MAGE based on the CGM data specified in the protocol
Percentage reduction in daily average of insulin use | 12 week, 24 week 52 weeks after transplant
  Change from baseline in insulin use specified in the protocol
Percentage of subjects with an HbA1c < 7.0 % assessed at 52 weeks post-transplant | One year after transplant
Percentage of subjects with an HbA1c ≤ 6.5 % assessed at 52 weeks post-transplant | One year after transplant
Percentage of subjects with positive porcine C-peptide qualitatively assessed by digital ELISA assay | One year after transplant
Values of porcine C-peptide during mixed meal tolerance test (MMTT) and Intravenous Glucose Tolerance Test (IVGTT) at each measuring point | For one year after transplant
  Assesment of glucose metabolism function
Psychological impact as assessed by the Diabetes Distress Scale (DDS) at each measuring point. | For one year after transplant
  Patient Quality of Life Assessment with DDS
Percentage of subjects with improved awareness of hypoglycemia, as defined by a change in Clarke questionnaire score from ≥ 4 to < 4. | For one year after transplant

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Hospital &Health Scences System, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No